CLINICAL TRIAL: NCT00909389
Title: Post - Marketing Surveillance of the Safety, Tolerability and Efficacy of Vytorin (Ezetimibe + Simvastatin) Tablet Among Filipino Patients
Brief Title: Post-marketing Surveillance of the Safety, Tolerability and Efficacy of Vytorin (Ezetimibe + Simvastatin) Tablet Among Filipino Patients (Study P05647)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05647
Record Dates: First submitted 2009-05-20; First posted 2009-05-28 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe; Simvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Filipino Patients with Hypercholesterolemia
  Interventions: Drug: Vytorin (R) (Ezetimibe + Simvastatin)

INTERVENTIONS:
Drug: Vytorin (R) (Ezetimibe + Simvastatin) — Vytorin (R) (Ezetimibe + Simvastatin) 1 tablet once daily to be taken by mouth in the evening for 28 days
  Other Names: SCH 465981

SUMMARY:
This study aims to establish the safety, tolerability, and efficacy of Vytorin (R) (Ezetimibe + Simvastatin) (SCH 465981) on a select population of Filipinos with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men or women, age 18 years and above
* Patients with primary (heterozygous familial and non-familial) hypercholesterolemia

Exclusion Criteria:

* Known hypersensitivity to Ezetimibe and Simvastatin
* Moderate to severe hepatic insufficiency
* Persistent elevation of serum transaminase levels of more than 1.5 times the upper limit of normal
* Pregnancy or lactation
* Concomitant intake of bile acid sequestrants (resins), nicotinic acid (niacin), fibric acid (fibrates), or cyclosporine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and above seen in the outpatient clinic who were diagnosed to have hypercholesterolemia. Patients with primary (heterozygous familial and non - familial) hypercholesterolemia or homozygous familial hypercholesterolemia were also included.
Sampling Method: Non-Probability Sample
Enrollment: 4748 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Filipino Patients With Hypercholesterolemia
Started | 4748
Completed | 4615
Not Completed | 133
Not completed — Adverse Event | 6
Not completed — Death | 4
Not completed — Poor Compliance | 16
Not completed — Lost to Follow-up | 4
Not completed — No Information | 103

BASELINE CHARACTERISTICS:
Arm/Group | Filipino Patients With Hypercholesterolemia
Number analyzed (Participants) | 4748
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.53 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2400
  Male | 2348

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had an Adverse Event (AE).
Description: The objective of this study was to evaluate the overall safety and tolerability of Vytorin (R) Tablet (Ezetimibe+Simvastatin) when used in patients with hypercholesterolemia.
  All AEs observed by or volunteered to the investigator during this observational study, regardless of suspected causal relationship, were to have been considered an AE.
Time Frame: Throughout study up to Day 29 (Final Visit)
Measure: Number; unit: participants
Arm/Group | Filipino Patients With Hypercholesterolemia
Number analyzed (Participants) | 4748
participants | 62

ADVERSE EVENTS:
Arm/Group | Filipino Patients With Hypercholesterolemia
Serious Adverse Events (participants affected / at risk) | 4/4748
Other Adverse Events (participants affected / at risk) | 0/4748
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filipino Patients With Hypercholesterolemia (N=4748)
Myocardial infarction (Cardiac disorders) | 1 (1) — Patient died.
Death (General disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1) — Patient died.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosures agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.